CLINICAL TRIAL: NCT01948999
Title: Electroconvulsive Therapy for Treatment Refractory Schizophrenia - A Randomized, Double-blinded, Sham-controlled Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Missing ressources. The study official has left and will not be replaced
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-20100085
Record Dates: First submitted 2013-06-17; First posted 2013-09-24 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Treatment-refractory Schizophrenia
Keywords: electroconvulsive therapy; treatment-refractory schizophrenia
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECT (Active Comparator): Electroconvulsive Therapy Anesthesia and concomitant muscular paralysis
  Interventions: Procedure: ECT; Drug: Anesthesia
- SHAM ECT (Sham Comparator): Anesthesia and concomitant muscular paralysis
  Interventions: Procedure: SHAM ECT; Drug: Anesthesia

INTERVENTIONS:
Procedure: ECT — Electroconvulsive Therapy inclusive anesthesia and concomitant muscular paralysis
  Arms: ECT
Procedure: SHAM ECT — Anesthesia and concomitant muscular paralysis
  Arms: SHAM ECT
Drug: Anesthesia — Temporary induced state of analgesia

SUMMARY:
The purpose of the study is to determine whether addition of electroconvulsive therapy to antipsychotic treatment improves the mental health of patients with treatment-resistant schizophrenia.

DETAILED DESCRIPTION:
The purpose of the study is not achieved.

ELIGIBILITY:
Inclusion Criteria:

* An ICD-10 schizophrenia diagnosis F20.0-20.3 or F20.9
* PANSS total score >= 70
* CGI-S >= 4 (Clinical Global Impression)
* PANSS score >= 4 on minimum 2 og the following items: Delusions, Conceptual disorganization,Hallucinatory behavior, Excitement, Grandiosity, Suspiciousness, Hostility, Disorientation.
* Previous/current treated with clozapine or refused clozapine treatment
* Lack of response to at least three different antipsychotics
* New antipsychotic medication prescribed more than 8 weeks before inclusion
* Fixed dosage of antipsychotics 1 month before inclusion
* No chance of additional neurotropic 4 weeks before inclusion
* Signed informed consent and power of attorney

Exclusion Criteria:

* Significant substance abuse
* Somatic disease that increases the risk of complications of ECT/anesthesia
* Epilepsy
* For women: Pregnancy or breast-feeding
* Homelessness
* Use of benzodiazepines (apart from tbl. oxazepam 10 mg., max 30 mg. daily)
* Use of antiepileptic
* Previous no effect on psychotic symptoms after ECT treatment (minimum 15 ECT- treatments)
* Concrete suicidal plans

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Reduction in total PANSS score and adverse events | The primary outcome will be assessed at screening, baseline and after every second week up to 72 weeks depending on the process for the individaul participant.
  PANSS = Positive and Negative Syndrome Scale and UKU = The UKU (Udvalg for Kliniske Undersøgelser) side effect rating scale

IPD SHARING:
Plan to Share IPD: No